CLINICAL TRIAL: NCT06219096
Title: Application of Indocyanine Green(ICG)@Human Serum Albumin(HSA) Complexes in Fluorescence Image-Guided Laparoscopic Anatomical Liver Resection: A Prospective, Double-Blinded, Randomized Controlled Trial
Brief Title: Application of ICG@HSA Complexes in Fluorescence Image-Guided Laparoscopic Anatomical Liver Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: Nanjing Chia-Tai Tianqing Pharmaceutical Company (Unknown)
Responsible Party: Principal Investigator, Hong Wu, Clinical Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IHLAP2121
Record Dates: First submitted 2023-12-25; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Malignant Tumor of Liver; Randomized Controlled Trial
Keywords: Indocyanine green; Laparoscopic anatomical hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study utilizes a double-blind design to ensure impartiality among operators, outcome assessors, and patients. The randomization assignment is only known to the research nurse, who administers the two different ICG administration protocols during surgery based on the assigned randomization number and group allocation. To maintain blinding, an opaque curtain is placed over the anesthesia operation area on the patient's head side, preventing the surgical operator from knowing the randomization assignment. The entire process of grouping and drug delivery is observed solely by the dedicated research nurse. In order to minimize assessment bias, the evaluators and data collectors are also blinded and have no knowledge of the patient's grouping information, thus reducing the potential impact of bias on the results. The efficacy of fluorescence imaging will be evaluated and scored independently by three experts in the field of fluorescence.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The new ICG & HSA injection Group (experimental group) (Experimental): After ligation of the targeted hepatic segmental portal vein, a novel ICG protocol is used (0.5mg ICG powder is added to 20mL normal saline containing 500mg human albumin, shaken and allowed to stand for more than 5 minutes to form a stable complex, with final concentrations of ICG 0.025mg/mL and human albumin 25mg/mL). This ICG-albumin conjugate solution is then administered intravenously at a rate of 1mL/min. The infusion is stopped when sufficient fluorescence enhancement is observed in the negative-staining liver regions.
  Interventions: Procedure: NIF image-guided laparoscopic anatomical liver resection with the novel ICG@HSA administration
- The guideline-recommended ICG injection Group (active comparator group) (Active Comparator): After ligation of the targeted hepatic segmental portal vein, 2.5mg of ICG (concentration 2.5mg/mL) is administered intravenously as a bolus injection.
  Interventions: Procedure: NIF image-guided laparoscopic anatomical liver resection with the guideline-recommended ICG administration

INTERVENTIONS:
Procedure: NIF image-guided laparoscopic anatomical liver resection with the novel ICG@HSA administration — After ligation of the target hepatic segmental portal vein, the novel ICG regimen (0.5 mg ICG powder and 500 mg human serum albumin added to 20 ml saline, shaken and allowed to stand for more than 5 minutes, ICG: 0.025 mg/ml, human serum albumin: 25 mg/ml) was intravenously infused continuously at a rate of 1 ml/min until significant fluorescence imaging appeared in the demarcated area, upon which the infusion was terminated.
  Arms: The new ICG & HSA injection Group (experimental group)
Procedure: NIF image-guided laparoscopic anatomical liver resection with the guideline-recommended ICG administration — After ligation of the target hepatic segmental portal vein, 2.5 mg of ICG (2.5 mg/ml) was intravenously injected.
  Arms: The guideline-recommended ICG injection Group (active comparator group)

SUMMARY:
This study is a single-center, prospective, randomized controlled trial that aims to compare the efficacy and safety of a new indocyanine green (ICG) administration protocol with the current guideline-recommended protocol for near-infrared (NIR) fluorescence imaging in laparoscopic anatomical hepatic resection. Primary liver cancer is a common malignancy worldwide. Laparoscopic liver resection has become increasingly popular due to its minimally invasive nature. During open and laparoscopic liver resection surgery, ICG, a fluorescent dye, is widely used to visualize liver segments and define tumor margins. However, there is a lack of high-level evidence regarding the timing and dosage of ICG administration in current protocols. In our preliminary study, we discovered a new method of pre-mixing ICG with albumin, which creates a more stable conjugate that could enhance fluorescence imaging during NIR laparoscopic hepatectomy. This study will include 100 patients with primary liver malignancies who are scheduled for laparoscopic anatomical hepatic resection. The patients will be randomly assigned in a 1:1 ratio to either the new ICG-albumin protocol (experimental group) or the standard ICG alone protocol (control group). The primary outcome will be the efficacy of fluorescence imaging, which will be evaluated using a 5-point scoring system by three independent experts. Secondary outcomes will include operation time, blood loss, tumor margin status, complications, length of stay, long-term recurrence, and survival.

The hypothesis of this study is that pre-binding ICG with albumin creates a more stabilized fluorescent complex, which could significantly improve the efficacy of fluorescence navigation and hepatectomy outcomes compared to standard ICG alone. This study aims to provide high-quality evidence on optimal protocols for ICG use in laparoscopic fluorescent image-guided liver surgery. The results of this study could help establish standardized guidelines to improve the application of this important navigation technique and enhance surgical precision and outcomes for liver cancer patients worldwide. The study protocol will be approved by the Ethics Review Board and publicly registered before enrollment starts. All participants will be required to provide informed consent. This study will be conducted in compliance with the Declaration of Helsinki and national regulations on human subject protection to ensure ethics, privacy, and safety.

DETAILED DESCRIPTION:
1. Study Design:

   This study is designed as a single center, prospective, randomized, double-blinded, controlled trial. The participants will be randomly assigned to either the experimental group (using the new ICG-albumin protocol) or the control group (using the standard ICG protocol) at a 1:1 ratio. The randomization will be done using a centralized web-based system.
2. Participants:

   The study aims to enroll 100 patients aged 18-75 years old with primary liver malignancies who are planned for laparoscopic anatomical hepatic resection at our institution. The main inclusion criteria are a Child-Pugh grade A or B liver function and an ECOG performance score of 0-1. The main exclusion criteria include an ICG R15 value of >=20%, coagulation disorders, severe heart/lung disease, active bleeding, allergy to ICG, severe gastroesophageal varices, and pregnancy/lactation.
3. Interventions:

   The interventions in the experimental group will involve mixing 0.5mg of ICG powder with 20mL saline containing 500mg of human albumin for at least 5 minutes. This mixture will then be intravenously infused at a rate of 1mL/min after occlusion of the target hepatic pedicles. On the other hand, the control group will receive a slow intravenous infusion of 2.5mg ICG (2.5mg/mL) following the current guidelines after pedicle occlusion.
4. Outcomes:

   The primary outcome is the efficacy of fluorescence imaging, which will be evaluated by a 5-point scoring system by three independent experts. Secondary outcomes include operation time, blood loss, conversion to open surgery, parenchymal transection time, use of hemostatic clips, tumor margins, postoperative complications, liver function recovery, length of stay, long-term recurrence and survival. Safety outcomes include complications, mortality, and adverse reactions associated with ICG.
5. Participant Timeline:

   Screening will take place within 2 weeks before surgery. Participants will be followed up during hospitalization. After discharge, follow-up will take place at month 1, 3, 6, 12, 18, 24, 30, 36 post-surgery.
6. Sample Size:

   With a two-sided 0.05 significance level, 90% power, and expecting a 1-point improvement in fluorescence imaging efficacy score (SD 1.5), 49 participants per group are needed, 100 in total.
7. Data Collection and Management:

   All data will be collected on paper case report forms and then entered into a centralized electronic data capture system. Data will go through quality check, cleaning, coding and logic validation. Any changes will be tracked. Cleaned and locked database will be used for final analysis. Original forms will be archived securely.
8. Statistical Analysis :

   Efficacy of fluorescence imaging will be compared between groups using t-test or Mann-Whitney U test. Operation parameters will be analyzed by t-test or Wilcoxon rank test. Tumor margins will be evaluated by chi-square test. Complication rates will be compared using t-test or Fisher's exact test. Survival outcomes will be depicted by Kaplan-Meier curves and compared by Log-rank tests. Multivariate Cox regression will be used to identify factors affecting recurrence and survival. Sensitivity analysis will be performed to account for missing data.
9. Data Monitoring:

   An independent data safety monitoring board will review study progress and safety data regularly. Any serious adverse events will be reported to investigators, IRB and regulatory agencies within 24 hours.
10. Ethics and Dissemination and Trial Status:

The study protocol will be approved by the IRB before initiation. All participants will provide written informed consent. Results will be disseminated through scientific conferences and peer-reviewed publications. The study is currently preparing for ethics submission and enrollment is expected to start in December 2023 and complete in November 2026.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old, patients with hepatic malignancies who are undergoing laparoscopic anatomical liver resection;
2. Preoperative liver function Child-Pugh grade A or B;
3. No contraindications for laparoscopic liver resection;
4. Expected survival ≥3 months;
5. ECOG PS score 0-1;
6. Normal major organ functions, and meet the following laboratory test results within 7 days prior to enrollment: white blood cell (WBC) ≥2.5×10^9/L, absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet (PLT) ≥75×10^9/L, hemoglobin (HGB) ≥90g/L; NR ≤1.5xULN; serum creatinine (CT) ≤1.5xULN; total bilirubin (TBI) ≤1.5×upper limit of normal (ULN);
7. Patients voluntarily participate and sign informed consent.

Exclusion Criteria:

1. No obvious ischemic demarcation line after intraoperative occlusion or disconnection of target hepatic pedicle, or the liver fluorescence reaches an intensity that interferes with surgery before intraoperative ICG injection.
2. Poor hepatic reserve function (ICG R15 ≥ 20%);
3. Severe cardiopulmonary diseases, intolerant to general anesthesia and surgery;
4. Moderate or large amount of symptomatic ascites or pleural effusion;
5. Active bleeding or coagulation abnormalities;
6. Hepatic encephalopathy;
7. Allergy to ICG;
8. History of gastrointestinal bleeding within the past 6 months or definite tendency for gastrointestinal bleeding;
9. Severe esophageal gastric varices requiring interventional treatment;
10. Objective evidence showing severe impaired pulmonary function such as pulmonary fibrosis;
11. Any significant clinical and laboratory abnormalities that the investigator considers affecting safety assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Fluorescence imaging effect of the live | On the 7th day after surgery
  The entire surgical video was recorded and then scored by experts

SECONDARY OUTCOMES:
Duration of surgery | At the end of the surgery
  Based on the duration of the surgery as recorded
Intraoperative bleeding | At the end of the surgery
  Based on the amount of bleeding recorded during the surgery
Conversion to laparotomy | At the end of the surgery
  Based on intraoperative records to determine whether to convert to open laparotomy
Duration of hepatic parenchymal transection | On the 7th day after surgery
  Organize a dedicated person to review the surgical video and record the duration after the surgery is over
Number of hemostatic clips used on the liver transection surface | On the 7th day after surgery
  Organize a dedicated person to review the surgical video and record the duration after the surgery is over
Tumor margins | At the end of the surgery
  Specimen tumor margins will be measured by pathologists using calipers
Postoperative complications | Up to 24 weeks after surgery
  Organize a dedicated person to record postoperative complications
Postoperative hepatic function | Up to 4 weeks after surgery
  Regularly measure liver function, coagulation, and other biochemical indicators after surgery after the patient returned to the ward
Postoperative bowel function recovery time | Up to 2 weeks after surgery
  Organize a dedicated person to record the time of rectal gas passage after surgery afer he patient returned to the ward
Postoperative hospital stay | On the second day after discharge
  Organize a dedicated person to record the postoperative hospital stay

OTHER OUTCOMES:
Overall survival | From date of randomization until death or loss to follow-up, up to 5 years
  Post-discharge follow-up (once every 3 months) using the follow-up center function of the professional EDC data management software to record follow-up via WeChat, questionnaires, and telephone calls
Disease-free survival | From the surgery was completed until disease progression or loss to follow-up, assessed up to 5 years
  Post-discharge follow-up (once every 3 months) using the follow-up center function of the professional EDC data management software to record follow-up via WeChat, questionnaires, and telephone calls

CONTACTS AND LOCATIONS:
Overall Officials: Hong Wu, Professor, Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Landsman ML, Kwant G, Mook GA, Zijlstra WG. Light-absorbing properties, stability, and spectral stabilization of indocyanine green. J Appl Physiol. 1976 Apr;40(4):575-83. doi: 10.1152/jappl.1976.40.4.575. PMID 776922
- [Result] Ishizawa T, Saiura A, Kokudo N. Clinical application of indocyanine green-fluorescence imaging during hepatectomy. Hepatobiliary Surg Nutr. 2016 Aug;5(4):322-8. doi: 10.21037/hbsn.2015.10.01. PMID 27500144
- [Result] Wang X, Teh CSC, Ishizawa T, Aoki T, Cavallucci D, Lee SY, Panganiban KM, Perini MV, Shah SR, Wang H, Xu Y, Suh KS, Kokudo N. Consensus Guidelines for the Use of Fluorescence Imaging in Hepatobiliary Surgery. Ann Surg. 2021 Jul 1;274(1):97-106. doi: 10.1097/SLA.0000000000004718. PMID 33351457
- [Result] Berardi G, Igarashi K, Li CJ, Ozaki T, Mishima K, Nakajima K, Honda M, Wakabayashi G. Parenchymal Sparing Anatomical Liver Resections With Full Laparoscopic Approach: Description of Technique and Short-term Results. Ann Surg. 2021 Apr 1;273(4):785-791. doi: 10.1097/SLA.0000000000003575. PMID 31460879
- [Result] Wakabayashi T, Cacciaguerra AB, Abe Y, Bona ED, Nicolini D, Mocchegiani F, Kabeshima Y, Vivarelli M, Wakabayashi G, Kitagawa Y. Indocyanine Green Fluorescence Navigation in Liver Surgery: A Systematic Review on Dose and Timing of Administration. Ann Surg. 2022 Jun 1;275(6):1025-1034. doi: 10.1097/SLA.0000000000005406. Epub 2022 Feb 2. PMID 35121701
- [Result] Chen H, Wang Y, Xie Z, Zhang L, Ge Y, Yu J, Zhang C, Jia W, Ma J, Liu W. Application Effect of ICG Fluorescence Real-Time Imaging Technology in Laparoscopic Hepatectomy. Front Oncol. 2022 Apr 6;12:819960. doi: 10.3389/fonc.2022.819960. eCollection 2022. PMID 35463377
- [Result] Itoh S, Tomiyama T, Morinaga A, Kurihara T, Nagao Y, Toshima T, Morita K, Harada N, Mori M, Yoshizumi T. Clinical effects of the use of the indocyanine green fluorescence imaging technique in laparoscopic partial liver resection. Ann Gastroenterol Surg. 2022 Mar 9;6(5):688-694. doi: 10.1002/ags3.12563. eCollection 2022 Sep. PMID 36091307
- [Result] Liu F, Wang H, Ma W, Li J, Liu Y, Tang S, Li K, Jiang P, Yang Z, He Y, Liu Z, Zhang Z, Yuan Y. Short- and Long-Term Outcomes of Indocyanine Green Fluorescence Navigation- Versus Conventional-Laparoscopic Hepatectomy for Hepatocellular Carcinoma: A Propensity Score-Matched, Retrospective, Cohort Study. Ann Surg Oncol. 2023 Apr;30(4):1991-2002. doi: 10.1245/s10434-022-13027-5. Epub 2023 Jan 16. PMID 36645540
- [Result] Cai X, Hong H, Pan W, Chen J, Jiang L, Du Q, Li G, Lin S, Chen Y. Does Using Indocyanine Green Fluorescence Imaging for Tumors Help in Determining the Safe Surgical Margin in Real-Time Navigation of Laparoscopic Hepatectomy? A Retrospective Study. Ann Surg Oncol. 2023 Apr;30(4):1981-1987. doi: 10.1245/s10434-022-12893-3. Epub 2022 Dec 9. PMID 36484905
- [Result] Xu Y, Chen M, Meng X, Lu P, Wang X, Zhang W, Luo Y, Duan W, Lu S, Wang H. Laparoscopic anatomical liver resection guided by real-time indocyanine green fluorescence imaging: experience and lessons learned from the initial series in a single center. Surg Endosc. 2020 Oct;34(10):4683-4691. doi: 10.1007/s00464-020-07691-5. Epub 2020 Jun 4. PMID 32500459
- [Derived] Xie Q, Gao F, Ran X, Zhao X, Yang M, Jiang K, Mao T, Yang J, Li K, Wu H. Application of indocyanine green-human serum albumin complex in fluorescence image-guided laparoscopic anatomical liver resection: study protocol for a randomized controlled trial. Trials. 2024 Dec 23;25(1):847. doi: 10.1186/s13063-024-08695-5. PMID 39710697